CLINICAL TRIAL: NCT03491683
Title: An Open-Label, Multi-Center Trial of INO-5401 and INO-9012 Delivered by Electroporation (EP) in Combination With REGN2810 in Subjects With Newly-Diagnosed Glioblastoma (GBM)
Brief Title: INO-5401 and INO-9012 Delivered by Electroporation (EP) in Combination With Cemiplimab (REGN2810) in Newly-Diagnosed Glioblastoma (GBM)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBM-001
Record Dates: First submitted 2018-04-02; First posted 2018-04-09 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; immunotherapy; DNA therapy; checkpoint inhibitor
MeSH Terms: conditions — Glioblastoma | interventions — rocakinogene sifuplasmid; cemiplimab; Radiotherapy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Cohort A: Unmethylated MGMT Promoter (Experimental): Cohort A will include participants with a glioblastoma tumor with an unmethylated MGMT promoter. Participants will receive INO-5401 and INO-9012 and cemiplimab as well as radiation and temozolomide (TMZ; only during radiation therapy), if clinically indicated.
  Interventions: Biological: INO-5401; Biological: INO-9012; Biological: Cemiplimab; Radiation: Radiation Therapy; Drug: Temozolomide
- Cohort B: Methylated MGMT Promoter (Experimental): Cohort B will include participants with a glioblastoma tumor with a methylated MGMT promoter or with indeterminate MGMT status. Participants will receive INO-5401 and INO-9012 and cemiplimab as well as radiation and temozolomide (TMZ), if clinically indicated. Participants will continue to receive TMZ following radiation therapy, for up to six additional cycles, if clinically indicated.
  Interventions: Biological: INO-5401; Biological: INO-9012; Biological: Cemiplimab; Radiation: Radiation Therapy; Drug: Temozolomide

INTERVENTIONS:
Biological: INO-5401 — INO-5401 is a combination of 3 separate DNA plasmids targeting Wilms tumor gene-1 (WT1) antigen, prostate-specific membrane antigen (PSMA) and human telomerase reverse transcriptase (hTERT) genes. Starting on Day 0 three milligrams (mg) of each plasmid will be delivered IM followed by EP using the CELLECTRA® 2000 EP device every three weeks for four doses, and then every 9 weeks until disease progression as defined by immunotherapy Response Assessment in Neuro-Oncology (iRANO), unacceptable toxicity, withdrawal of consent, or death.
Biological: INO-9012 — INO-9012 is a DNA plasmid for expression of human interleukin-12 (IL-12). Starting on Day 0 one mg plasmid will be delivered IM followed by EP using the CELLECTRA® 2000 EP device every three weeks for four doses, and then every 9 weeks until disease progression as defined by iRANO, unacceptable toxicity, withdrawal of consent, or death.
Biological: Cemiplimab — Cemiplimab is an antibody to programmed death-1 (PD-1) protein. Starting on Day 0 cemiplimab will be administered intravenously (IV) every three weeks at a dose of 350 mg per dose in the absence of dose holding, until disease progression as defined by iRANO, unacceptable toxicity, withdrawal of consent, or death.
  Other Names: REGN2810
Radiation: Radiation Therapy — Radiation therapy (RT) will begin no later than 42 days after surgical intervention, and should start approximately 2 weeks after Day 0. RT will be given for three weeks.
Drug: Temozolomide — Temozolomide (TMZ) will be given daily during radiation therapy (RT) at a dose of 75 milligrams per square meter (mg/m^2).

SUMMARY:
Phase 1/2 trial to evaluate safety, immunogenicity and preliminary efficacy of INO-5401 and INO-9012 in combination with cemiplimab (REGN2810), with radiation and chemotherapy, in subjects with newly-diagnosed glioblastoma (GBM).

DETAILED DESCRIPTION:
This is a phase 1/2, open-label, multi-center trial to evaluate safety, immunogenicity and preliminary efficacy of INO-5401 and INO-9012 in combination with cemiplimab in subjects with newly-diagnosed glioblastoma (GBM). INO-5401 and INO-9012 will be delivered by intramuscular (IM) injection followed by electroporation (EP) in combination with cemiplimab and chemoradiation and radiation. There will be 2 cohorts in this trial. Cohort A will be participants with a tumor with an unmethylated O6-methylguanine-deoxyribonucleic acid (DNA) methyltransferase (MGMT) promoter. Cohort B will be participants with a tumor with a MGMT methylated promoter or who have indeterminate MGMT status. Both cohorts will receive INO-5401 and INO-9012 and cemiplimab at the same doses and on the same dosing schedule, and both cohorts will receive radiation and temozolomide (TMZ), if clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Newly-diagnosed brain cancer with histopathological diagnosis of GBM;
* Karnofsky Performance Status (KPS) rating of >/=70 at baseline;
* Receive dexamethasone equivalent dose </=2 mg per day, stable or decreased for >/= three days prior to Day 0;
* Recovery from the effects of prior GBM surgery as defined by the Investigator;
* Electrocardiogram (ECG) with no clinically significant findings as assessed by the Investigator;
* Adequate organ function as demonstrated by hematological, renal, hepatic laboratory assessments;
* Agree that during the trial, men will not father a child, and women cannot be or become pregnant. Participants must be of non-child bearing potential or agree to use one highly effective or combined contraceptive methods that result in a failure rate of <1% per year during the treatment period and at least through week 12 after last dose;
* Ability to tolerate magnetic resonance imaging (MRI).

Exclusion Criteria:

* Presence of greater than 1 cm x 1 cm residual tumor enhancement on postoperative MRI;
* Multifocal disease or leptomeningeal disease (LM) disease on post-operative MRI;
* Not scheduled to start radiation within 42 days of surgical resection of tumor;
* Dexamethasone equivalent dose >2 mg per day;
* Prior treatment with an agent that blocks the PD-1/PD-Ligand 1 pathway;
* Receipt of previous approved or investigative immune modulatory agent within 28 days of receiving the first dose of treatment;
* Prior treatment with idelalisib;
* Past, current or planned treatment with tumor treatment fields; oncolytic viral treatment; or prior exposure to an investigational agent or device within 28 days of receiving the first dose of treatment;
* Allergy or hypersensitivity to cemiplimab or to any of its excipients;
* History of documented allergic reactions or acute hypersensitivity reaction attributed to antibody treatments;
* Ongoing or recent (within 5 years) evidence of autoimmune disease that required treatment with systemic immunosuppressive treatments;
* Diagnosis of immunodeficiency or treatment with systemic immunosuppressive therapy within 28 days prior to the first dose of trial treatment, other than dexamethasone for the underlying disease under investigation, as noted in the inclusion criteria;
* History of clinically significant, medically unstable disease which, in the judgment of the investigator, would jeopardize the safety of the subject, interfere with trial assessments or endpoint evaluation, or otherwise impact the validity of the trial results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | From Day 0 to 30 days after the last dose of study treatment (non-serious AEs) and to 6 months after the last dose of study treatment (immune-related AEs, AEs of special interest and serious AEs) up to approximately 24 months

SECONDARY OUTCOMES:
Overall survival at 18 months (OS18) | At Month 18
Change from Baseline in Interferon-gamma Secreting T Lymphocytes in Peripheral Blood Mononuclear Cells (PBMCs) | From Day 0 to last dose of study treatment up to approximately 18 months
Change from Baseline in T-Cell Phenotypes in PBMCs | From Day 0 to last dose of study treatment up to approximately 18 months
Change from Baseline in T Cell Receptor (TCR) Subtypes in PBMCs | From Day 0 to last dose of study treatment up to approximately 18 months
Change from Baseline in Antigen-Specific Humoral Response | From Day 0 to last dose of study treatment up to approximately 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Skolnik, MD, Study Director — Inovio Pharmaceuticals
Locations (21):
- United States (21):
  - City of Hope, Duarte, California
  - Stanford University, School of Medicine, Palo Alto, California
  - University of California, San Francisco, San Francisco, California
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Rutgers University - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New York University Langone Medical Center; Perlmutter Cancer Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center The Neurological Institute of New York, New York, New York
  - New York-Presbyterian Hospital/Weill Cornell Medical Center, New York, New York
  - University of North Carolina School of Medicine, Chapel Hill, North Carolina
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania Health System: Penn Medicine, Philadelphia, Pennsylvania
  - UPMC Cancer Center Neuro-Oncology; UPMC Cancer Pavilion, Pittsburgh, Pennsylvania
  - Texas Oncology, Austin, Texas
  - Baylor College of Medicine, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah